CLINICAL TRIAL: NCT04316598
Title: Monocenter, Double-Blind, Randomized, Placebo-Controlled, Parallel Group Study to Assess the Pharmacodynamic Effects of Cannabis on Neural Oscillations in Healthy Recreational Cannabis Users
Brief Title: Cannabis Effects on Electroencephalography
Acronym: CEG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by the sponsor in the context of COVID-19 pandemia
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IMIMFTCL_CEG
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
Keywords: Cannabis; Recreational drugs; Neural oscillations; THC
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, double-blind, randomized, placebo-controlled, parallel group study. Subjects will be randomly assigned in a 2:1 ratio to study arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The subjects, Investigators and designees involved in the conduct of the study will be blinded to the identity of the treatment administered during the study.
  The following precautions will be taken to ensure the integrity of the study blinding during the trial:
  * The monodose capsules containing the treatment conditions will be prepared by an unblinded technician who will not be involved in any study assessment. The unblinded technician will also maintain records for drug accountability.
  * Treatment will not be unblinded for an individual subject except for a medical emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabis (B) (Experimental): Subjects will be admitted in the center to receive 4 doses of inhaled cannabis in 3 days.
  Vital signs, blood test and electroencephalogram (Starlab® helmet) will be performed before and after every cannabis administration. Cannabis subjective effects will be assessed and a psychiatric research interview will also be performed at different times after administration.
  Interventions: Drug: Cannabis Sativa
- Cannabis placebo (B) (Placebo Comparator): Subjects will be admitted in the center to receive 4 doses of an inhaled treatment based on placebo-THC in 3 days.
  Vital signs, blood test and electroencephalogram (Starlab® helmet) will be performed before and after every administration. Cannabis subjective effects will be assessed and a psychiatric research interview will also be performed at different times after administration.
  Interventions: Drug: Cannabis placebo

INTERVENTIONS:
Drug: Cannabis Sativa — Subjects will receive a total of 4 inhaled doses of 20 mg of tetrahydrocannabinol (THC) in 3 days.
  Cannabis is provided as a medical grade cannabis flos (Cannabis sativa dried female flower) containing THC 22% and cannabidiol <1%, supplied by Bedrocan®.
  To avoid the respiratory disadvantages of smoking, a vaporization device (Mighty® Medic) will be used to inhale the drug. The prepared capsules will contain 90 mg of Cannabis flos, equivalent to 20 mg of THC.
  Other Names: THC; Bedrocan®
  Arms: Cannabis (B)
Drug: Cannabis placebo — Subjects will receive a total of 4 inhaled doses of cannabis placebo (THC <0,2%) in 3 days.
  Placebo cannabis is provided as a medical grade cannabis flos (Cannabis sativa dried female flower) containing cannabinoids <0.2%. To avoid the respiratory disadvantages of smoking, a vaporization device (Mighty® Medic) will be used to inhale the drug. The prepared capsules will contain 90 mg of cannabis placebo.
  Other Names: Knaster
  Arms: Cannabis placebo (B)

SUMMARY:
Background:

Tetrahydrocannabinol (THC) is a partial CB1/CB2 agonist and causes its pharmacological effects by binding to cannabinoid receptors. CB1 receptors are predominantly located in the brain (highest densities at hippocampus, cerebellum and the striatum) and at low levels in the brainstem. CB2 receptors are predominantly in the spleen and in hematopoietic cells. THC is highly lipophilic and is readily absorbed and distributed to the brain and other organs.

Most of the neuropsychological studies carried out so far show that the mainly affected neurocognitive functions in cannabis users are: memory, attention, psychomotor capacity, speed of information processing and alterations of executive functions (resistance to interference, planning capacity, decision-making, verbal fluency and working memory). These effects are dose-dependent.

Hypothesis:

Functional CB1 receptor activation by the THC contained in the cannabis flos will induce dose-dependent effects on EEG, physiological functions and behavior:

1. EEG alterations.
2. Increase in cannabis subjective effects.
3. Increase in heart rate.
4. Increase in psychopathology scale Psychotomimetic State Inventory (PSI) score.
5. Increase in plasma cortisol concentrations.

Objectives:

Main pharmacodynamic objective: To assess the effects of Cannabis flos on electroencephalography (EEG) in healthy recreational cannabis users.

Secondary pharmacodynamic objectives: (i) To assess the effects of Cannabis flos on: cannabis subjective effects, heart rate and psychopathology scale; (ii) To establish the pharmacokinetic/pharmacodynamic relationships between THC plasma concentrations and pharmacodynamic endpoints.

Safety and tolerability objectives: To assess the safety and tolerability of THC in these subjects.

Methods:

Phase I, prospective, monocentric, double-blind, randomized, placebo-controlled, parallel group study to assess the THC effects on EEG neural oscillations in 16 healthy subjects with recreational cannabis use.

DETAILED DESCRIPTION:
Subjects will be randomly assigned in a 2:1 ratio to either Arm A (Cannabis) or Arm B (Cannabis placebo). The subjects, Investigators and designees involved in the conduct of the study will be blinded to the identity of the treatment administered during the study.

In the active group (Arm A) subjects will be administered four single doses of 20 mg THC over 3 days, equivalent to 285.7 μg/kg. This dose is considered to be sufficient for eliciting the psychoactive effects of THC (> 5 ng/mL in plasma) and modify EEG, avoiding subjects to be too much behaviorally impaired.

THC will be administered in the form of medical cannabis (Bedrocan®) inhaled by intrapulmonary route. It is featured in flos form (Cannabis sativa dried female flower) containing THC 22% and cannabidiol (CBD) <1%. A vaporization system (Mighty® Medic device) will be used for cannabis administration. Through this system, the final inhalation of THC is comparable to that of smoking cannabis while reducing the inhalation of toxic and irritating substances generated in the combustion of herbs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects.
* Negative urine pregnancy test and effective contraception method for female of child-bearing potential (see footnote at the end of subheading 5).
* Age ≥ 18 and ≤ 55 years.
* Weight ≥ 50 kg and ≤ 100 kg.
* Body mass index (BMI) ≥ 18 and ≤ 30.
* Recreational cannabis use with a cannabis use history ≥ 6 months and a cannabis consumption in the last month ≥ 1 day/month and ≤ 2 days/week.
* Last cannabis consumption ≥ 1 week before Day 1.
* Negative urine drug test but for cannabis.
* Consistent drug hair test (performed during screening) with drug use medical history.
* Able to read Spanish and adhere to study requirements.
* Not under any administrative or legal supervision.
* Signed informed consent prior to any study-mandated procedure.

Exclusion Criteria:

* Pregnant or nursing female.
* Cannabis-naive subjects.
* Life-time cannabis use disorder (CUD) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria using the Psychiatric Research Interview for Substance and Mental Disorders (PRISM).
* Recreational use of opioids, cocaine, psychostimulants within the last month.
* Life-time other substance use disorders (SUD) according to the DSM-5 criteria using PRISM, except for mild alcohol use disorder and/or mild or moderate nicotine use disorder.
* Life-time history of bipolar disorders, psychosis or suicidal attempts assessed by the Dual Diagnosis Screening Instrument (DDSI).
* Past-12 months history of anxiety or depression assessed by the DDSI.
* Life-time clinically significant cardiovascular, renal, pulmonary, hepatic, onco-hematological, endocrine, gastrointestinal or neurological disease.
* Any other diseases or conditions that in the judgment of the investigator would interfere with the subject's ability to comply with study procedures or requirements and/or study results interpretation.
* Any clinically significant findings in physical examination including vital signs, EEG and safety laboratory parameters.
* Any prescription or over the counter drug (except occasional use of paracetamol) in the last 2 weeks before Day 1 of each period.
* Patient included in a clinical study in the last three months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with EEG alterations | 45 minutes pre-administration to 45 minutes post-administration
  THC induced EEG alterations, such as:
  * Decrease in phase synchronization (intertrial coherence) of the 40 Hertz gamma band assessed by the auditory steady state response (ASSR).
  * Decrease in evoked power of the 40 Hertz gamma band assessed by the auditory steady state response (ASSR).
  * Decrease in P300 wave amplitude assessed by a three-stimulus auditory oddball task.
  * Decrease in power of neural oscillations in resting state eyes-closed EEG.
  * Increase in EEG complexity, measured by the Lempel-Ziv complexity.
  * Decrease in EEG brain connectivity (band coherence, synchronicity likelihood) in resting state eyes-closed/open.
  * Decrease in cross-frequency theta-gamma coupling.

SECONDARY OUTCOMES:
Number of Participants with subjective effects | Before administration, at 15, 50, 75 and 105 minutes post-administration
  THC induced alterations in subjective and psychotomimetic effects, measured as increase in cannabis subjective effects and increase in psychopathology scale Psychotomimetic State Inventory (PSI) score.
Number of Participants with alterations in cardiovascular function | Before administration to 60 minutes post-administration
  THC induced alterations in cardiovascular function, such as increased heart rate measured by a wearable medical device.
Number of Participants with neuroendocrine alterations | Before administration, at 10 and 60 minutes post-administration
  THC induced neuroendocrine alterations, such as increased cortisol plasma concentrations.
Time-profile of THC | Before administration, at 10 and 60 minutes post-administration
  Changes in concentration of THC in blood
Time-profile of OH-THC | Before administration, at 10 and 60 minutes post-administration
  Changes in concentration of OH-THC in blood
Time-profile of THC-COOH | Before administration, at 10 and 60 minutes post-administration
  Changes in concentration of THC-COOH in blood

CONTACTS AND LOCATIONS:
Overall Officials: Rafael de la Torre Fornell, Dr, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No